CLINICAL TRIAL: NCT03911297
Title: Dissecting Androgen Excess and Metabolic Dysfunction for an Integrated Systems Approach to Polycystic Ovary Syndrome Through the Assessment of Detailed Phenome and Metabolome Data
Brief Title: DAISy-PCOS Phenome Study - Dissecting Androgen Excess and Metabolic Dysfunction in Polycystic Ovary Syndrome
Acronym: DAISy-PCOS
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: University Hospital Birmingham NHS Foundation Trust (Other); Birmingham Women's and Children's NHS Foundation Trust (Other); University Hospital of Wales (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); Royal Infirmary of Edinburgh (Other); Royal College of Surgeons, Ireland (Other); Imperial College Healthcare NHS Trust (Other); Hull University Teaching Hospitals NHS Trust (Other Government); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19HH5264; WT209492/Z/17/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2019-04-08; First posted 2019-04-11 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; androgens; steroids; metabolic risk; prediction; stratified medicine
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be stored in a Human tissue act approved site and ethics for a potential future analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Women with polycystic ovary syndrome — Prospective cohort study in women with polycystic ovary syndrome to identify the risk of developing metabolic disease

SUMMARY:
Polycystic ovary syndrome (PCOS) affects 10% of all women and usually presents with irregular menstrual periods and difficulties conceiving. However, PCOS is also a lifelong metabolic disorder and affected women have an increased risk of type 2 diabetes, high blood pressure, and heart disease. Increased blood levels of male hormones, also termed androgens, are found in most PCOS patients. Androgen excess appears to impair the ability of the body to respond to the sugar-regulating hormone insulin (=insulin resistance). The investigator has found that fat tissue of PCOS patients overproduces androgens and that this can result in a build-up of toxic fat, which increases insulin resistance and could cause liver damage. In a large cohort of women registered in a GP database, the study team have found that androgen excess increases the risk of fatty liver disease. The aim is to identify those women with PCOS who are at the highest risk of developing metabolic disease, which would allow for early detection and potentially prevention of type 2 diabetes, high blood pressure, fatty liver and cardiovascular disease. The investigator will assess clinical presentation, androgen production and metabolic function in women with PCOS to use similarities and differences in these parameters for the identification of subsets (=clusters) of women who are at the highest risk of metabolic disease. The investigator will do this by using a standardised set of questions to scope PCOS-related signs and symptoms and the patient's medical history and measure body composition and blood pressure. This standardised recording of a patient's clinical presentation (=clinical phenotype) is called Phenome analysis. The investigator will collect blood and urine samples for the systematic measurement of steroid hormones including a very detailed androgen profile (=steroid metabolome analysis) and of thousands of substances produced by human metabolism (=global metabolome analysis). Phenome and metabolome data will then undergo integrated computational analysis for the detection of clusters predictive of metabolic risk.

DETAILED DESCRIPTION:
The investigator propose an innovative approach to solving the clinical problem at hand, the lack of identified measurable parameters one can use to predict the risk of future metabolic disease in women diagnosed with PCOS.The chosen approach is the standardised collection of phenome and metabolome data and their unbiased integration by machine learning analysis. Utilising the detailed results of the clinical phenome and metabolome analysis in the DAISy-PCOS Phenome Study cohort, The study will aim to identify distinct subsets (=clusters) of PCOS patients that share similar characteristics. This approach has previously been used by the team to successfully identify distinct steroid markers that can serve as a "malignant steroid fingerprint" in urine to distinguish benign from malignant tumours in patients with incidentally discovered adrenal masses. Similarly, The investigator have used unbiased analysis of steroid metabolome data to reveal that patients with aldosterone excess also overproduce glucocorticoids and that the latter explains the majority of metabolic disease risk observed in affected patients.

In the integrated analysis of the DAISy-PCOS phenome and metabolome data, The investigator will apply a variety of methods in the context of connectivity or centroid-based clustering and density estimation. Supervised relevance learning will give insight into markers, e.g. steroids, that are most decisive for the determination of cluster memberships. In addition, The investigator will use state-of-the-art visualisation and machine learning techniques based on adaptive similarity measures.the investigator will use integrative approaches, addressing the heterogeneous data from different sources as a whole, whilst considering data-driven adaptation of generative models for the underlying biological processes. The investigator will employ these approaches to characterise central phenotype clusters affecting large numbers of patients as the basis of personalised management including outcome prediction.

ELIGIBILITY:
Inclusion Criteria:

* Women with a suspected diagnosis of polycystic ovary syndrome
* Age range 18-70 years
* Ability to provide informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding at the time of planned recruitment
* History of significant renal (eGFR<30) or hepatic impairment (AST or ALT >two-fold above ULN; pre-existing bilirubinaemia >1.2 ULN)
* Any other significant disease or disorder that, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participants who have participated in another research study involving an investigational medicinal product in the 12 weeks preceding the planned recruitment
* Glucocorticoid use via any route within the last six months
* Current intake of drugs known to impact upon steroid or metabolic function or intake of such drugs during the six months preceding the planned recruitment
* Use of oral or transdermal hormonal contraception in the three months preceding the planned recruitment
* Use of contraceptive implants in the twelve months preceding the planned recruitment

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women with a new diagnosis of Polycystic ovary syndrome aged 18-70 who are treatment naive
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic risk | 5 years
  Metabolic-risk prediction model would be made from a machine learning algorithm where the study team would be able to enter phenome and metabolome data of patient with a new diagnosis of PCOS. With this model, the study team would be able to stratify the women with PCOS into their risk of metabolic disease hence personalise the management of the condition

SECONDARY OUTCOMES:
Dissect the severity and pattern of androgen excess in development of metabolic disease | 5 years
  The study team would assess how pattern of androgen excess in each phenotype relates to their risk of metabolic disease
Eligibility for other PCOS-related studies | 3 years
  Participants will be screened for their eligibility to enroll in other PCOS-related research studies

CONTACTS AND LOCATIONS:
Overall Officials: Wiebke Arlt, Principal Investigator — University of Birmingham
Locations (1):
- Wellcome Trust Clinical Research Facility, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No